CLINICAL TRIAL: NCT00079820
Title: The Safety, Tolerability, and Immunogenicity of Three Dose Levels of ACAM3000 Modified Vaccinia Ankara (MVA) Smallpox Vaccine, in Adults Without Previous Smallpox Vaccination
Brief Title: Safety, Tolerability, and Immune Response of ACAM3000 Modified Vaccinia Ankara (MVA) Smallpox Vaccine in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-249-001
Record Dates: First submitted 2004-03-15; First posted 2004-03-17 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Smallpox
Keywords: Smallpox; Smallpox Vaccine; Variola virus; Smallpox Virus; MODIFIED VACCINIA ANKARA; MVA; Dryvax; Dryvax vaccine; Protection against smallpox
MeSH Terms: conditions — Smallpox | interventions — DryVax vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- A (Experimental): MVA3000 Smallpox vaccine (1x10-8) with Dryvax Challenge at Day 112
  Interventions: Biological: ACAM3000 MVA Vaccine
- B (Experimental): MVA3000 Smallpox vaccine (1x10-8) with no Challenge
  Interventions: Biological: ACAM3000 MVA Vaccine
- C (Placebo Comparator): Placebo
  Interventions: Biological: ACAM3000 MVA Vaccine
- D (Experimental): MVA3000 Smallpox vaccine (1x10-7) with Dryvax challenge at Day 112
  Interventions: Biological: ACAM3000 MVA Vaccine
- E (Experimental): MVA3000 Smallpox vaccine (1x10-6) with Dryvax challenge at Day 112
  Interventions: Biological: ACAM3000 MVA Vaccine

INTERVENTIONS:
Biological: ACAM3000 MVA Vaccine — Two subcutaneous injections of MVA3000 smallpox vaccine, separated by 28 days
  Other Names: Dryvax smallpox vaccine

SUMMARY:
The purpose of this study is to gather information on the safety and the effectiveness of an investigational vaccine for the prevention of smallpox disease. Smallpox was one of the major causes of death and sickness through the first half of the 20th century, but a global program of smallpox eradication resulted in the elimination of the natural disease. The last cases of smallpox in the United States occurred in 1949 in Texas. Today, only laboratory workers who work with smallpox-related viruses, military personnel, and health care workers are vaccinated.

Historically, individuals in the US were vaccinated with a product such as Dryvax®, which contains the virus vaccinia in the same family as smallpox. This virus could promote immunity to smallpox, but not produce the disease itself. Although effective, these vaccines are not safe to use in people with atopic dermatitis (eczema, allergic immune response to allergens), children less than 1 year of age, and people with a compromised immune system, occurring in certain diseases (HIV positive individuals and AIDS), and following treatment with certain types of drugs. It is important to find a safe vaccine that can be used to protect people who cannot receive routine vaccinia-based smallpox vaccine.

The vaccine in this study is known as Modified Vaccinia Ankara or MVA vaccine. It is the objective of this study to find out if MVA vaccine is safe and effective in providing immunity to smallpox. The effectiveness of this vaccine will be measured in two ways. The first way is to find out if there are specific antibodies in your blood following MVA vaccination. Antibodies are chemicals your body produces to fight smallpox virus.

The second way is to see whether or not there is a typical skin reaction following vaccination with a traditional smallpox vaccine, given about three months after vaccination with the MVA vaccine. The typical reaction in an unvaccinated person to smallpox vaccine is formation of a blister or "pox" which occurs at the site of vaccination. In a person with immunity to smallpox the skin reaction is much less, and typically consists of a little swelling at the site of vaccination.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following to be eligible for the study:

* adult males or females who provided informed consent for the study.
* adults 18 and 31 years (inclusive).
* good general health,
* female subjects must not be pregnant or lactating and be on appropriate contraception or be a female unable to bear children.
* subjects be available for participation during the entire study.

Exclusion Criteria:

Any of the following exclusion criteria are met, the subject is NOT eligible.

* military service prior to 1989 or after December 13th, 2002.
* history of previous smallpox vaccination
* known/suspected history of immunodeficiency, or with current radiation treatment or use of immunosuppressive or anti-neoplastic drugs.
* subjects with a household member or intimate contact with the same conditions listed above.
* known or suspected impairment of other immunologic function.
* malignancy, including squamous cell or basal cell skin cancer at vaccination site
* active autoimmune disease.
* subjects with known eye diseases or other conditions that require the use of corticosteroid eye drops.
* known/history of cardiac disease.
* subjects who have been diagnosed with 3 or more of the following risk factors for ischemic coronary disease: a) high blood pressure b) elevated blood cholesterol levels c) diabetes or high blood sugar d) first degree relative (for example, mother, father, brother, or sister) who had a heart condition before the age of 50 e) smoke cigarettes
* subjects with a history of palpitations or abnormalities of cardiac rhythm.
* subjects with odd ECG patterns
* subjects with a ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years.
* positive or elevated creatinine kinase, CK-MB, or Troponin I laboratory test levels.
* abnormalities of clinical laboratory assessments.
* past history or current diagnosis of chronic renal disease, adverse reactions to drugs characterized by renal impairment, a serum creatinine > 1.5 mg/dL, or presence of 1+ protein in urinalysis at screening and a calculated creatinine clearance of not less than 80 mL/min.
* current diagnosis or past history of eczema.
* subjects with a household member or intimate contact with the same conditions listed above.
* presence of acute, chronic, or exfoliative skin conditions, open wounds, or burns.
* history of keloid formation.
* known allergies to MVA or to any known components (Neomycin, Gentamycin) of the vaccine.
* known allergy to eggs or egg products.
* known allergies to any component of the Dryvax® vaccine. Antibiotics in Dryvax® include neomycin, streptomycin, chlortetracycline, and polymixin B.
* known allergies to any known component of the Dryvax® diluent (i.e., glycerin and phenol).
* known allergies to any known component of VIG, (i.e., thimerosal or previous allergic reaction to immunoglobulins).
* known allergies to cidofovir or sulphur containing drugs, including probenecid, trimethoprim, and sulfonamide antibiotics.
* transfusion of blood or treatment with any blood product, including intramuscular or intravenous serum globulin within 6 months of the screening visit.
* positive serology result for HIV, hepatitis B surface antigen, or hepatitis C.
* current diagnosis or history within six months of the screening visit of drug or alcohol abuse disorders.
* significant acute or chronic psychiatric illness.
* female subjects with a positive serum pregnancy test result
* subjects with a household member or direct contact with someone who is pregnant or lactating.
* temperature or acute illness within 3 days prior to vaccination
* inoculation with an inactivated vaccine with 14 days of Day 0 or with a live attenuated vaccine within 30 days of Day 0.
* subjects who have participated in another investigational drug or vaccine trial within 30 days of Day 0.
* subjects who are planning on donating blood or organs within 30 days of vaccination.

Ages: 18 Years to 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2004-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Safety | Study Completion

SECONDARY OUTCOMES:
Immunogenicity | Study Completion

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (2):
- United States (2):
  - PRA International, Lenexa, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky